CLINICAL TRIAL: NCT04407195
Title: Mental Health Outcomes Among US Healthcare Workers Exposed to COVID-19
Brief Title: COVID-19 and Mental Health
Status: Completed | Type: Observational
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Kara Pavone, Assistant Professor, Northeastern University
Other Study IDs: 20-05-22
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: COVID-19; Mental Health Disorder
MeSH Terms: conditions — COVID-19; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Providers: Healthcare workers (physicians and nurses) who have interacted with patients with known or suspected COVID-19.
  Interventions: Other: Exposure to the SARS-CoV-2

INTERVENTIONS:
Other: Exposure to the SARS-CoV-2 — This is an observational design. Participants are exposed to the Covid-19 pandemic.

SUMMARY:
The overall objective of this study is to assess the enormity of mental health outcomes among healthcare providers (nurses and physicians) exposed to COVID-19 during the time of the pandemic in the United States, specifically targeting those areas most effected.

DETAILED DESCRIPTION:
Healthcare providers (nurses and physicians) on the frontlines of the COVID-19 response are facing a critical situation and are subject to increased psychological distress. Those directly involved in the diagnosis, treatment and care of patients with COVID-19 are at significant risk of developing physical, psychological, and psychosocial distress.

The data examined in this study will further clarify the mental distress experienced by healthcare workers and lead to the development of peer-support and educational initiatives to improve these findings. The central hypothesis of this research is that high levels of mental distress will be associated with caring for patients with COVID-19.

This study will use an observational, cross-sectional on-line survey design. Participants will complete a 15 minute self-administered questionnaire. All data will be de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers (physicians and nurse) working in institutions with known or suspected COVID-19.

Exclusion Criteria:

* Nurses and physicians who are retired, or not currently employed or not working in an environment with known or suspected COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include physicians and nurse who interact with patients with known or suspected COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Emotional Impact | 7 days
  The Impact of Event Scale - Revised (IES-R). IES-R is a 22-item scale with possible scores ranging from 0 - 88. Scores higher than 24 are of concern indicating possible health and well-being consequences.

SECONDARY OUTCOMES:
Depression | 2 weeks
  Patient Health Questionaire (PHQ-9). The PHQ-9 has a range from 0 - 27. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression.
Anxiety | 2 weeks
  Generalized Anxiety Disorder 7-item (GAD-7). Scores range from 0 - 21. When screening for anxiety disorders, a score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder.
Insomnia | 1 week
  The ISI7 is a 7-item instrument designed to assess the nature, severity, and impact of insomnia in adults. Scores range from 0 - 28. Higher scores indicate increased likelihood of sleep disturbances.
Resilience | 2 Weeks
  Brief Resilience Scale (BRS) is a 6-item scale with scores ranging from 6-30 with higher scores indicating greater resilience.
Crisis Support Scale | 2 weeks
  The Crisis Support Scale (CSS) is a 7-item instrument developed to measure received social support. Scores range from 7 - 98, with higher scores correlating with increased social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No